CLINICAL TRIAL: NCT00643981
Title: Phase I Study to See if a of A Combination Stem Cell Therapy is Safe and Feasible for the Treatment of Severe Coronary Ischemia
Brief Title: Combination Stem Cell Therapy for the Treatment of Severe Coronary Ischemia
Acronym: CI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Gabriel P. Lasala, M.D., TCA Cellular Therapy, LLC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-03-I
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2008-12

CONDITIONS: Coronary Ischemia; Coronary Disease; Coronary Artery Disease; Coronary Atherosclerosis; Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

INTERVENTIONS:
Biological: MESENDO — 2 ml of the "final cell mixture" will be injected through the lumen of an intracoronary percutaneous balloon designed for angioplasty into the ishcemic vessel.

SUMMARY:
The purpose of this research study is to determine if the infusion of a combination of stem cells obtained from the bone marrow of the same patient will contribute to the formation of new blood vessels in patients with symptomatic severe coronary ischemia. In this trial we will study the safe use of this therapy and its effects on making new blood vessels will be evaluated.

Coronary ischemia is intractable angina due to severe coronary artery disease which can seriously decrease blood flow to the heart.

CI needs a comprehensive treatment since the condition will not improve on its own. The overall goal of the treatment is to increase blood flow to the heart and improve symptoms of angina.

The study hypothesis is based on the concept that the process of formation of new blood vessels is complex and requires the participation of several types of stem cells and growth factors. The lack of any of these components will produce vessels which are immature and unable to provide appropriate blood supply to the heart.

Patients eligible to participate in this study are those suffering from severe blockages to the vessels of the heart and are not candidates for percutaneous revascularization or surgical procedures.

Once the final mixture of stem cells is prepared, the cells will be intracoronary infused through a catheter into the blocked vessel of the heart.

Studies will be performed to evaluate if the intracoronary infusion of stem cells is safe, feasible and works.

Patients will be evaluated for 6 months after cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18-20
* Angina Pectoris: CCS Class II or IV or angina symptom equivalent
* 70% blockage in at least one epicardial vessel documented within 6 months
* Stable medical therapy
* Reversible perfusion defects by SPECT
* Not a candidate for percutaneous intervention or coronary by-pass surgery

Exclusion Criteria:

* Previous angiogenic therapy or myocardial laser therapy
* Severe valvular heart disease
* Recent malignancy or radiation therapy within 6 months
* Renal insufficiency with creatinine greater that 2.7
* White blood count greater than 13,000 or lower than 3,000
* Platelet count lower than 60,000 or higher that 500,000
* Pregnant or planning to become pregnant
* History of skeletal muscle disease
* AST or ALT greater than two times upper limit of normal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety as measured by laboratory assessments, ecg, temperature and holter monitor | 2 weeks

SECONDARY OUTCOMES:
Efficacy as measured by SPECT scan and 2-D Echo | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- TCA Cellular Therapy, LLC, Covington, Louisiana, United States